CLINICAL TRIAL: NCT06957548
Title: Screening for Cardiometabolic Disease Risk Factors: a Community Health Screening Program in Urban Cameroon
Brief Title: Cardiometabolic Disease Risk Factors in Cameroon
Acronym: URBACAM-D
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00474444
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Disease; Metabolic Disease
MeSH Terms: conditions — Heart Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiometabolic disease — Cardiometabolic disease screening

SUMMARY:
Cardiometabolic diseases (CMDs) are a major public health concern in sub-Saharan Africa, including Cameroon. Studies have shown a significant increase in the prevalence of hypertension, diabetes, and obesity in recent years. However, access to timely diagnosis and treatment remains limited, particularly in rural areas. Community-based screening programs have been shown to be effective in identifying individuals with undiagnosed CMD risk factors and promoting early intervention. By leveraging the strengths of community-based approaches, the URBACAM-D study aims to address the growing burden of CMDs in urban Cameroon.

ELIGIBILITY:
Inclusion Criteria:

* Screening is open to any adult over the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urban Cameroon. Newbell, Douala, cameroon.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2025-10-12 (Actual); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Cardiometabolic disease risk factors in Urban Cameroon | 1 year
  To determine the prevalence of undiagnosed and uncontrolled cardiometabolic disease (CMD) risk factors among urban Cameroonians.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Tito, DO, Principal Investigator — Johns Hopkins University
Locations (1):
- Newbell Protestant Hospital, Douala, Littoral Region, Cameroon